CLINICAL TRIAL: NCT01455064
Title: FreeStyle Navigator II Continuous Glucose Monitor Home Use Evaluation (FSNv2)
Brief Title: Navigator II Continuous Glucose Monitor Home Use Study
Status: Completed | Type: Observational
Sponsor: Abbott Diabetes Care (Industry)
Responsible Party: Sponsor
Other Study IDs: ADC11-106
Record Dates: First submitted 2011-10-15; First posted 2011-10-19 (Estimated); Results first posted 2013-07-22 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-05

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Type 1 or 2 diabetes, MDI or pump
  Interventions: Device: FreeStyle Navigator II Continuous Glucose Monitoring System

INTERVENTIONS:
Device: FreeStyle Navigator II Continuous Glucose Monitoring System — This is not an interventional study. Subjects must maintain their own diabetes treatment regimen throughout the study duration

SUMMARY:
This research study will test a new investigational continuous glucose monitoring system (System). The purpose of this study is to find out about the performance of the System in a home use environment over a 15 day period, in people with diabetes.

ELIGIBILITY:
Inclusion Criteria:

The subject must:

* Have type 1 or 2 diabetes for at least 2 years prior to enrollment.
* Require insulin therapy administered through an insulin pump or multiple daily injections (MDI) for at least 6 months prior to enrollment.
* Be at least 18 years of age.
* Be able to read and understand English.
* In the investigator's opinion, be able to follow the instructions provided to him/her by the study site and perform all study tasks as specified by the protocol.
* Be available for all study visits.
* Be willing to provide written signed and dated informed consent.

Exclusion Criteria:

The subject must not:

* Be pregnant or likely to become pregnant during the study duration.
* Have skin abnormalities at the insertion sites.
* Have known allergy to medical grade adhesive or skin disinfectant.
* Be using a continuous glucose monitor currently or within the past 6 months
* Have a concomitant medical condition which, in the opinion of the investigator, could interfere with the study or present a risk to the safety or welfare of the subject.
* Be participating in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 1 or 2 diabetes requiring multiple daily insulin injections or using an insulin pump
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2011-10; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shridhara A Karinka, Ph.D., Study Director — Abbott Diabetes Care
Locations (2):
- United States (2):
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Southwest Clinical Research Center, Santa Fe, New Mexico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from within the patient population of two US diabetes clinical centers.
Groups:
- Observational Group: Participants using the FreeStyle Navigator II RT-CGM for 15 days (360 hours).
Period: Overall Study
Arm/Group | Observational Group
Started | 31
Completed | 30
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Observational Group
Number analyzed (Participants) | 31
Age, Customized [Mean (Full Range); unit: years] | 48.4 [21 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 16
Weight [Mean (Full Range); unit: kilograms] | 90.4 [52.6 to 163.7]
Height [Mean (Full Range); unit: meters] | 1.70 [1.50 to 1.93]
Years since diagnosis [Mean (Full Range); unit: years] | 19.6 [5 to 47]
Daily total insulin dosage [Mean (Full Range); unit: units] | 72.8 [22 to 186]
Total number of injections per day [Mean (Full Range); unit: injections (N subjects = 18)] | 3.6 [2 to 5]

OUTCOME MEASURES:

1. Primary Outcome: Clarke Error Grid Analysis
Description: Percentage of CGM results in the clinically accurate Zone A and percentage of CGM results in the clinically acceptable Zones A and B of the Clarke Error Grid versus blood glucose reference.
Time Frame: 15 days sensor wear
Population: One subject was withdrawn due to a mild reaction to the sensor adhesive. This subject's data was included in the study up to the point of withdrawal.
Measure: Number; unit: Percentage of Results
Units Other Than Participants: Results
Arm/Group | Observational Group
Number analyzed (Participants) | 31
Number analyzed (Results) | 2843
Percentage of Results
  Percentage of results in Clarke Error Zone A | 83.0
  Percentage_Results in Clarke Error Zones A&B | 97.7

ADVERSE EVENTS:
Arm/Group | Observational Group
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 4/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Observational Group (N=31)
Severe hypoglycemia (Endocrine disorders) | 1 (1) — Not device related, Not procedure related, Severity = Severe, non-serious adverse event, unanticipated
Scabbing (Skin and subcutaneous tissue disorders) | 2 (2) — Device-related, procedure-related, severity = moderate, non-serious adverse event, anticipated. Device-related, procedure-related, severity = mild, non-serious adverse event, anticipated.
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) — Device-related, procedure-related, severity = mild, non-serious adverse event, anticipated
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) — Device-related, procedure-related, severity = mild, non-serious adverse event, anticipated
Laryngitis (General disorders) | 1 (1) — Not device related, not procedure related, severity = moderate, non-serious adverse event, unanticipated
Ear infection in right ear (Infections and infestations) | 1 (1) — Not device related, not procedure related, severity = moderate, non-serious adverse event, unanticipated

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days